CLINICAL TRIAL: NCT03939585
Title: Preemptive Infusion of Donor Lymphocytes Depleted of TCR (Alpha-beta) + T Cells and CD19+ B Cells Following Allogeneic Stem Cell Transplantation
Brief Title: Preemptive Infusion of Donor Lymphocytes Depleted of TCR + T Cells + CD19+ B Cells Following ASCT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Leland Metheny (Other)
Responsible Party: Sponsor-Investigator, Leland Metheny, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1Z19
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Allogeneic Stem Cell Transplant Candidate; Acute Myeloid/Lymphoblastic Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Lymphoproliferative Disorders
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoproliferative Disorders

STUDY DESIGN:
Intervention Model Description: This is a Phase I, pilot study designed to treat 10 participants with the donor NK/γδ T cell-enriched product on transplant Day 28.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NK/γδ T cell-enriched cell therapy product (Experimental): This study will treat 10 participants with the donor NK/TCR-γδ T cell product. Of those 10 participants, 5 would have 10/10 HLA matched sibling donors (MSD) while 5 would have partially matched, related (haplo) donors.
  * 27 days post transplant, the participant's donor will undergo a second, non-mobilized leukapheresis to obtain peripheral blood mononuclear cells (PBMCs).
  * Donor PBMCs will be processed next day (Day T+28) to obtain the NK cell/TCRγδ T cell product for same day infusion if the participant remains aGVHD free and clinically stable.
  * Participants will continue routine post-transplant and GVHD monitoring, as well as disease assessment at 56 days, 100 days, 6 months and 1 year following transplant.
  * Blood samples will be obtained on T=0, T+7, 14, 21 and 28 days and then weekly until T + 56 days, then on T+100 days, + 6 months and + 12 months. If immune-mediated adverse events occur (GVHD, CRS etc) additional blood samples will be obtained at onset and resolution.
  Interventions: Biological: Cellular therapy product

INTERVENTIONS:
Biological: Cellular therapy product — Cellular therapy product: Allogeneic transplant donor lymphocytes, depleted of TCR-αβ T cells and B cells; enriched for NK cells and TCRγδ T cells.
  * Infused using venous catheter on post-transplant Day 28 (+ 7 days).
  * Single infusion of entire lymphocyte product derived from two-blood volume leukapheresis (non-mobilized).

SUMMARY:
The purpose of this study is to reduce the risk of cancer relapse by giving a donor lymphocyte infusion (DLI) to boost the immune system early after a stem cell transplant so that leukemia cells that escaped chemotherapy can be detected and killed. This DLI will contain mostly lymphocytes that have graft versus tumor effect with low risk of graft versus host disease. Because the process of giving a DLI in the first four weeks after a transplant has not been approved by the Food and Drug Administration (FDA), this study in investigational (experimental).

DETAILED DESCRIPTION:
The primary objective of this study is to investigate if donor lymphocytes depleted of TCR-αβ T cells and B cells can be infused on Day 28 following allogeneic stem cell transplantation without inducing Grade III-IV graft versus host disease, Grade II GVHD requiring systemic treatment and or new onset, severe neutropenia requiring growth factor support.

This study also seeks to characterize the lymphocyte subsets obtained following depletion of TCR-αβ T cells and B cells from non-mobilized, leukapheresis products.

Additionally, this study will attempt to describe occurrence of disease relapse and to describe the occurrence of post-transplant re- activation and/or infections with viruses such as CMV, and EBV.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologic or cytologic confirmation of ANY hematologic malignancy
* Allogeneic stem cell transplant is indicated as management of underlying hematologic malignancy.
* Participant has organ function (cardiac, lung and liver) considered adequate to undergo conditioning chemotherapy and allogeneic stem cell transplant in the assessment of the clinical program
* Participant has a 10/10 HLA-matched sibling donor OR has a HLA-haploidentical donor available (in the absence of a 10/10 HLA matched unrelated donor)
* The related transplant donor is willing, available and consents to undergo a second, non-mobilized leukapheresis for the procurement of donor lymphocytes
* The related transplant donor is 18 years of age or older
* Subjects must have the ability to understand and the willingness to sign a written informed consent document or provide assent.

Exclusion Criteria:

* Subject is unwilling to receive a prophylactic donor lymphocyte infusion per study protocol.
* The related donor is unwilling or unavailable to undergo a second, non- mobilized leukapheresis for the procurement of donor lymphocytes.
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 4 weeks prior to study entry and for the duration of study participation. Women of child-bearing age must have documented negative pregnancy test prior to start of conditioning regimen for stem cell transplantation and a repeat negative pregnancy test prior to infusion of the lymphocyte product.
* Patients with any of the following organ function abnormalities: Left ventricular ejection fraction (LVEF) < 45%; DLCO <45% of expected value corrected for alveolar volume and hemoglobin; Serum Creatinine >2 times the upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade III-IV GVHD, Grade II GVHD requiring systemic treatment or new onset, severe neutropenia requiring growth factor support at Day 100 and T+6 months. | up to 30 days after lymphocyte product infusion
  This study seeks to measure if donor lymphocytes depleted of TCR-αβ T cells and B cells can be infused on Day 28 following allogeneic stem cell transplantation without inducing Grade III-IV graft versus host disease, Grade II GVHD requiring systemic treatment or new onset, severe neutropenia requiring growth factor support.
  The endpoint associated with this objective is 'incidence of Grade III-IV graft versus host disease, Grade II GVHD requiring systemic treatment or new onset, severe neutropenia requiring growth factor support at Day 100 and T+6 months.'

SECONDARY OUTCOMES:
Different lymphocyte types in the infused product reported as cells per kilogram body weight of the recipient | 28 days post-transplant
  Number of different lymphocyte types in the infused product measured as cells per kilogram body weight of the recipient
Number of disease relapse events in the first 6 moths following stem cell transplant | 6 months from start of treatment
  To describe occurrence of disease relapse, the number of disease relapse events in the first year following stem cell transplant will be reported.
Number of disease relapse events in the first 1 year following stem cell transplant | 1 year from start of treatment
  To describe occurrence of disease relapse, the number of disease relapse events in the first year following stem cell transplant will be reported.
Average time to disease relapse from date of transplant | 6 months from start of treatment
  To describe occurrence of disease relapse, the average time to disease relapse from date of transplant in the first six months following stem cell transplant will be reported.
Average time to disease relapse from date of transplant | 1 year from start of treatment
  To describe occurrence of disease relapse, the average time to disease relapse from date of transplant in the first year following stem cell transplant will be reported.
Occurrence of reactivated Epstein Barr Virus (EBV) and/or Cytomegalovirus viremia (CMV) as measured by number of study subjects developing measurable viremia | 6 months from start of treatment
  To describe the occurrence of post-transplant re- activation and/or infections with viruses such as CMV, and/or EBV, the number of study subjects developing measurable viremia will be reported
Average time to first occurrence of reactivated EBV and/or CMV | 6 months from start of treatment
  To describe the occurence of post-transplant re- activation and/or infections with viruses such as CMV, and/or EBV, median time to first occurrence of reactivated EBV and/or CMV will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Leland Metheny, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie or influence the results observed from the study
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Investigators who provide a methodologically sound proposal for use of requested data